CLINICAL TRIAL: NCT05142904
Title: Ultrasound-guided Radiofrequency Ablation Versus Radioactive Iodine as Treatment for Hyperthyroidism Caused by Solitary Autonomous Thyroid Nodules
Brief Title: Radiofrequency Ablation Versus I-131 for Solitary Autonomous Thyroid Nodules
Acronym: RABITO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Switched from RCT to observational prospective cohort due to termination of subsidy (delay due to insufficient inclusion-rate). Follow-up of RCT-arm will be completed. Patients can still be included in a observational cohort.
Sponsor: Rijnstate Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); University of Twente (Other); Amsterdam UMC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1798
Record Dates: First submitted 2021-11-05; First posted 2021-12-03 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Nodule, Toxic or With Hyperthyroidism; Autonomous Thyroid Function; Thyroid Nodule; Hyperthyroidism; Radiofrequency Ablation; Iodine Hyperthyroidism; Iodine Adverse Reaction
MeSH Terms: conditions — Thyroid Nodule; Hyperthyroidism | interventions — Radiofrequency Ablation; Transurethral Resection of Prostate; Iodine-131

STUDY DESIGN:
Intervention Model Description: Multicentre 1:1 randomized clinical trial where patients are allocated to either radiofrequency ablation (RFA) or radioactive iodine (RAI) (I-131). Patients who are not suitable for randomization (e.g. no informed consent or contra-indication for RFA) are asked for consent to participate in a prospective cohort where participants are asked to fill out questionaires and data is collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radiofrequency ablation (Experimental): Patients allocated to the radiofrequency ablation (RFA) arm will undergo RFA under local anaesthesia with the moving-shot technique.
  Interventions: Device: Radiofrequency ablation
- Radioactive iodine, study protocol (Active Comparator): Patients allocated to this arm will undergo treatment with radioactive iodine (I-131) according to a standardized dose-calculation.
  Interventions: Drug: Radioactive iodine
- Radioactive iodine, cohort (Other): This group contains patients who are not randomized and have given informed consent undergo treatment with radioactive iodine (I-131) according to local standard (e.g. fixed dose or dose-calculation based on iodine uptake and thyroid nodule mass).
  Interventions: Drug: Radioactive iodine

INTERVENTIONS:
Device: Radiofrequency ablation — Ultrasound-guided radiofrequency ablation of the solitary autonomous thyroid nodule.
  Other Names: RFA; Ultrasound-guided radiofrequency ablation
  Arms: Radiofrequency ablation
Drug: Radioactive iodine — I-131 according to standardized doses-calculation.
  Other Names: I-131
  Arms: Radioactive iodine, study protocol
Drug: Radioactive iodine — I-131 according to local standard.
  Other Names: I-131
  Arms: Radioactive iodine, cohort

SUMMARY:
The purpose of this study is to compare treatment of hyperthyroidism with radiofrequency ablation or I-131 for solitary autonomous thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hyperthyroidism or subclinical hyperthyroidism caused by a solitary hyperactive thyroid nodule (HTN), either located in an otherwise normal thyroid gland, or in a multinodular goitre (MNG), with a diagnosis based on the following characteristics:

  * Blood TSH level below the lower limit of normal, and associated with either normal or elevated FT4 and FT3 levels
  * Anti-TSH antibody negative
  * Solitary HTN confirmed by a diagnostic I-123 scintigraphy, corresponding with a well demarcated thyroid node on ultrasound, cystic degeneration < 75%, nodule size <50 mm.
* Treatment with RAI indicated, and eligible for RFA treatment
* Signed informed consent Patients who are ineligible for randomization due to unsuitability for RFA, may be eligible for the RAI cohort group.

Exclusion Criteria:

* Multifocal HTN
* HTN > 50 mm
* Presence of a medical device susceptible to disturbances caused by RFA generated currents
* Patients with physical or behavioural disorders that preclude safe isolation in radiation protection rooms, or safe RFA procedure under local anesthesia
* Patients with dysphagia, oesophageal stenosis, active gastritis, gastric erosion, a peptic ulcer or impaired gastro-intestinal motility
* Uncorrectable haemorrhagic diathesis
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Hypothyroidism | 1 year post-intervention
  Incidence of hypothyroidism (defined as TSH above normal values with/without decreased FT4 and/or FT3 levels)

SECONDARY OUTCOMES:
Cure rate | 1 year post-intervention
  Medication-free normalization of TSH, FT4 and FT3 levels
Thyroid nodule volume | Baseline, 6 and 12 months post-intervention
  Volume of thyroid nodule assessed by ultrasound
Treatment related adverse events | 6 weeks and 3, 6 and 12 months post-intervention
  Number of adverse and serious adverse events
Thyroid related quality of life | Baseline, 6 and 12 months after intervention
  Thyroid related quality of life assessed by ThyPro questionnaire
Cost-effectiveness | Baseline, 6 weeks, and 3, 6, 9 and 12 months post-intervention
  Determined as the incremental costs in Euros per quality adjusted life year (QALY)
Course of thyroid function | Baseline, 1 and 6 weeks, 3, 6, 9 and 12 months post-intervention with an extension of follow-up up to 5 years.
  Assessed by TSH, FT4 and FT3 an medication use
Short-term patient satisfaction | 1 week and 1 year post-intervention
  Assessed by interviews, satisfaction questionnaire and pain scoring by visual analog scale (VAS, a scale ranging from 0-10 represented as a line with 0 on the left end indicating 'no pain' and 10 on the right end, indicating 'the worst pain').

OTHER OUTCOMES:
Health outcomes and quality of life | Baseline, 6 and 12 months after intervention
  Assessed by European Quality of Life-5 Dimensions (EQ-5D) questionnaire. ( questions in 5 dimensions with 3 response levels, a higher score representing a worse outcome)
Use of hospital resources | 1 year post-intervention
  According to medical records
Medical consumption | 1 year post-intervention
  iMCQuestionnaire (institute for medical technology assessment medical consumption questionnaire)
Use of healthcare resources | 1 year post-intervention
  iPCQuestionnaire (institute for medical technology assessment productivity cost questionnaire)
Cumulative cost | 1 year post-intervention
  Based on Rijnstate price estimates
Fractional nodal uptake | 1 year post-intervention
  Assessed by I-123 or I-131 scintigraphy
Treatment related auto-immunity | Baseline and 1 year post-intervention
  Assessed by thyroid antibodies

CONTACTS AND LOCATIONS:
Locations (14):
- Netherlands (14):
  - Ziekenhuis Groep Twente, Almelo, Gelderland
  - Gelre Hospitals, Apeldoorn, Gelderland
  - Rijnstate Hospital, Arnhem, Gelderland
  - Laurentius Hospital, Roermond, Limburg
  - Amphia Hospital, Breda, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - Elkerliek Hospital, Helmond, North Brabant
  - Amsterdam UMC, location VUMC, Amsterdam, North Holland
  - OLVG, Amsterdam, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Albert Schweiter Hospital, Dordrecht, South Holland
  - Haaglanden MC, The Hague, South Holland
  - Haga Ziekenhuizen, Zoetermeer, South Holland
  - Martini Hospital, Groningen

IPD SHARING:
Plan to Share IPD: No